CLINICAL TRIAL: NCT00520169
Title: A Randomized, Open Label, Single Center, Single-Dose, Cross-Over Study to Determine the Absolute Bioavailability and the Nasopharyngeal Absorption of PMI-150 (Intranasal Ketamine) in Healthy Adult Volunteers
Brief Title: Absolute Bioavailability and Nasopharyngeal Absorption of Intranasal Ketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KET-PK-007
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): oral ketamine
  Interventions: Drug: intranasal ketamine
- B (Experimental): intranasal ketamine
  Interventions: Drug: intranasal ketamine
- C (Active Comparator): intravenous ketamine
  Interventions: Drug: intranasal ketamine

INTERVENTIONS:
Drug: intranasal ketamine — A randomized, open label, single center, single-dose study to determine the absolute bioavailability and nasopharyngeal absorption of PMI-150 (intranasal ketamine) 30mg in healthy adult volunteers. The Pilot Phase will be conducted as a parallel study, while the Test Phase will be conducted as a crossover study.

SUMMARY:
This is an open label, single-center study to determine the absolute bioavailability and nasopharyngeal absorption of PMI-150 (intranasal ketamine) 30 mg in healthy adult volunteers.

DETAILED DESCRIPTION:
To examine the safety and assess the absolute bioavailability and nasopharyngeal absorption of PMI-150 30mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
ketamine pharmacokinetics | multiple

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmaceuticals
Locations (1):
- Javelin Pharmaceuticals, Cambridge, Massachusetts, United States